CLINICAL TRIAL: NCT01354444
Title: Pilot Trial of Carvedilol in Alzheimer's Disease
Brief Title: Trial of Carvedilol in Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00035546
Record Dates: First submitted 2011-05-09; First posted 2011-05-16 (Estimated); Results first posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Alzheimer's Disease
Keywords: Memory problems; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease; Memory Disorders | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carvedilol (Active Comparator): Carvedilol is a is a beta-blocker. Beta-blockers are generally used to reduce the workload on the heart and help it to beat more regularly.
  Interventions: Drug: Carvedilol
- Placebo (Placebo Comparator): Non active substance
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carvedilol — target dose of 25 mg daily which is half the maximum dose used in clinical practice
  Arms: Carvedilol
Drug: Placebo — a pill that will look like the active drug but will not contain any carvedilol
  Arms: Placebo

SUMMARY:
This is a 6-month pilot randomized double-blind placebo-controlled trial of carvedilol, with the primary objective being to determine whether carvedilol treatment is associated with improvement in Alzheimer's Disease (AD) as compared to placebo treatment. Secondary objectives are to monitor changes in cerebrospinal fluid amyloid levels and whether this dose will be safe and well-tolerated in AD patients. Clinical assessments will be performed at baseline, 3 months, and 6 months, while cerebrospinal fluid and blood samples will be obtained at baseline and 6 months.

DETAILED DESCRIPTION:
The purpose of the study is to measure decline in episodic memory in participants with early AD taking carvedilol compared to placebo treatment as evidenced by the Hopkins Verbal Learning Test (HVLT). cerebrospinal fluid levels of Aβ oligomers in early AD, will be measured in participants receiving carvedilol treatment when compared to placebo treatment. Adverse effects will be monitored in participants receiving carvedilol when compared to placebo.

To assess adverse events, routine chemistry and hematology studies, vital signs, and electrocardiographic parameters before and after 6 months randomized placebo-controlled double-blind treatment with carvedilol at a target dose of 25 mg daily, comparing 25 early AD participants taking carvedilol vs. 25 early AD participants taking placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD by the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria
* Mini-Mental State Exam (MMSE) 16-26. This range corresponds roughly to "mild" AD as rated by CDR below, and provides a rapid test for efficient screening of potential participants.
* Clinical Dementia Rating (CDR) < 1 (mild dementia). This corresponds with "early" AD. Participants will be eligible if they have AD diagnosis and CDR of 0.5 or 1.0. The category of CDR 0.5 AD is particularly important to include as these participants are in the earliest stage that can be diagnosed as dementia (as opposed to mild cognitive impairment) and thus are in the "earliest" clinical stage of AD.
* Patients will be allowed to remain on current FDA-approved Alzheimer's treatments including cholinesterase inhibitors and memantine, so long as the dose has been stable for >= 3 months. These medications lack any notable effects on amyloid synthesis or metabolism and thus there is no reason to exclude them. The rationale behind requiring a stable dose is so that change in the trial can be attributed to the study intervention rather than recent changes of other medications affecting cognition.
* Patients will be allowed to remain on antidepressant and antipsychotics medications so long as the dose has been stable for >= 3 months. The rationale is the same as above.
* Knowledgeable informant available for all study visits. This is standard practice in AD research because many standard instruments and questionnaires in this trial require a knowledgeable informant.

Exclusion criteria

* Evidence of non-AD dementias including Huntington's disease, Parkinson's disease, or frontotemporal dementia.

  2.Current Diagnostic and Statistical Manual Diploma in Social Medicine (DSM)-IV Axis I diagnoses other than dementia, including major depression, bipolar disorder, schizophrenia, anxiety disorders, alcohol abuse, or other substance abuse. These diagnoses would merit their own treatment plans and changes in these conditions could significantly affect cognitive and functional outcomes, confounding our efforts to study the efficacy of the study intervention.
* Any clinically significant medical condition that could interfere with the subject's ability to safely participate in the study or to be followed.
* Current use of Beta-blocking agents.
* Contraindications to use of Beta-blocking agents, to be determined in consultation with the patient's primary care physician or (if appropriate) cardiologist.
* Clinically significant hepatic or renal insufficiency.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul B. Rosenberg, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine Bayview Campus, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carvedilol | Placebo
Started | 14 | 15
Completed | 6 | 11
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carvedilol | Placebo | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 9 | 9 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 4 | 9 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 11 | 14 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Hopkins Verbal Learning Test (HVLT) Scores at Baseline, 3, and 6 Months
Description: The investigators measured episodic memory (as evidence by the Hopkins Verbal Learning Test (HVLT)) before and after 6 months randomized placebo-controlled double-blind treatment with carvedilol at a target dose of 25 mg daily. Changes in HVLT Immediate and Delayed Recall score in 14 Alzheimer's Disease (AD) participants taking carvedilol vs. 15 AD participants taking placebo were compared. HVLT test score ranges are as follows: immediate recall (0-24) delayed recall (0-12). Higher scores indicate better episodic memory recall.
Time Frame: Baseline, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- HVLT Score in Placebo Group: Descriptive statistics for immediate recall in the Hopkins Verbal Learning Test in the placebo group
- HVLT Score in Treatment Group: Descriptive statistics for immediate recall in the Hopkins Verbal Learning Test in the treatment group
Arm/Group | HVLT Score in Placebo Group | HVLT Score in Treatment Group
Number analyzed (Participants) | 15 | 14
Scores on a scale
  HVLT score at Baseline (immediate recall) | 13 (4) | 12 (6)
  HVLT score at 3 months (immediate recall) | 12 (5) | 13 (4)
  HVLT score at 6 months (immediate recall) | 12 (5) | 13 (6)
  HVLT score at Baseline (delayed recall) | 1 (2) | 1 (1)
  HVLT score at 3 months (delayed recall) | 1 (2) | 1 (2)
  HVLT score at 6 months (delayed recall) | 1 (2) | 0 (0)
Statistical Analysis 1: Comparison: HVLT Score in Placebo Group vs HVLT Score in Treatment Group; This analysis compares immediate recall before and after 6 months between the treatment and placebo group; Test type: Other; p = 0.565, Regression, Linear; Coefficient = 1.48, 95% CI 2-sided [-3.796 to 6.761]

2. Secondary Outcome: Effect of Carvedilol Treatment in Cerebrospinal Fluid (CSF) Levels of Amyloid-beta Oligomers
Description: The investigators will measure CSF Abeta oligomer levels before and after 6 months randomized placebo-controlled double-blind treatment with carvedilol at a target dose of 25 mg daily, comparing the change in levels in 6 AD participants taking carvedilol vs. 10 AD participants taking placebo. These 16 participants had both baseline and 6 month CSF collected (of the entire study population). CSF was collected at the baseline visit and 6 months later.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Carvedilol | Placebo
Number analyzed (Participants) | 6 | 10
pg/mL
  Baseline Tau (pg/mL) | 169.476 (93.931) | 169.484 (48.386)
  Baseline ABeta42 (pg/mL) | 396.985 (212.411) | 379.406 (100.892)
  Baseline P tau (pg/mL) | 42.666 (10.176) | 66.133 (24.503)
  Six month Tau (pg/mL) | 222.461 (139.839) | 171.757 (53.72)
  Six month ABeta42 (pg/mL) | 499.325 (174.308) | 361.563 (89.044)
  Six month P tau (pg/mL) | 56.003 (23.984) | 64.331 (25.766)
Statistical Analysis 1: Comparison: Carvedilol vs Placebo; This analysis compares the change in total Tau between the treatment and placebo group from baseline to 6 months later; Test type: Other; p = 0.481, Rank sum test
Statistical Analysis 2: Comparison: Carvedilol vs Placebo; This analysis compares the change in Abeta42 between the treatment and placebo group from baseline to 6 months later; Test type: Other; p = 0.0562, Rank sum test
Statistical Analysis 3: Comparison: Carvedilol vs Placebo; This analysis compares the change in p-tau between the treatment and placebo group from baseline to 6 months later; Test type: Other; p = 0.314, Rank sum test
Statistical Analysis 4: Comparison: Carvedilol vs Placebo; This analysis compares the change in oligomeric Abeta between the treatment and placebo group from baseline to 6 months later; Test type: Other; p = 0.438, Rank sum test

3. Secondary Outcome: Effect of Carvedilol Treatment in Cerebrospinal Fluid (CSF) Levels of Amyloid-beta Oligomers
Description: The investigators will measure CSF Abeta oligomer levels before and after 6 months randomized placebo-controlled double-blind treatment with carvedilol at a target dose of 25 mg daily, comparing the change in levels in 6 AD participants taking carvedilol vs. 10 AD participants taking placebo. These 16 participants had both baseline and 6 month CSF collected (of the entire study population).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Carvedilol | Placebo
Number analyzed (Participants) | 6 | 10
ng/mL
  Baseline Oligomeric ABeta (ng/mL) | 3.83 (3.314) | 0.129 (0.034)
  Six month oligomeric ABeta (ng/mL) | 3.895 (3.376) | 0.117 (0.101)

ADVERSE EVENTS:
Description: Adverse Events are presented without regard to the specific Adverse Event Term.
Arm/Group | Carvedilol | Placebo
Serious Adverse Events (participants affected / at risk) | 2/14 | 1/15
Other Adverse Events (participants affected / at risk) | 12/14 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carvedilol (N=14) | Placebo (N=15)
HEME (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
GI (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neurologic (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carvedilol (N=14) | Placebo (N=15)
HEME (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cardiac (Cardiac disorders) | 10 (10) | 10 (10)
Systemic (Nervous system disorders) | 2 (2) | 4 (4)
Dermatologic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psychiatric (Psychiatric disorders) | 1 (1) | 5 (5)
GI (Gastrointestinal disorders) | 2 (2) | 3 (3)
Neurologic (Nervous system disorders) | 2 (2) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Infectious disease (Infections and infestations) | 1 (1) | 1 (1)
Oncology (Immune system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes